CLINICAL TRIAL: NCT05761340
Title: The Effect of Helfer Skin Tap Technique on Pain Reduction and Hemodynamic Parameters During Tetanus Injection in Pregnant Women
Brief Title: The Effect of Helfer Skin Tap Technique During Tetanus Injection in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Celal Bayar University
Record Dates: First submitted 2023-01-25; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Intramuscular Injection; Pain
Keywords: Intramuscular Injection; Pain; Helfer Skin Tap Technique; Hemodynamic parameters
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: Pregnant women meeting the inclusion criteria were assigned to the Helfer skin tap and standard application groups by a computer-based random number generator. The numbers in set 1 were taken to the Helfer skin tap group and the numbers in set 2 to the standard application group by lot method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Helfer Skin Tap Group (Experimental): Pregnant women were vaccinated against tetanus with the Helfer skin tap technique.The pain was evaluated with Number rating scale immediately after the procedure and also hemodynamic parameters were measured before and after the vaccination. A total of 33 pregnant women completed the study in the Helfer skin tap group
  Interventions: Procedure: Helfer skin tap injection technique
- Standard Application Group (Experimental): Pregnant women were vaccinated against tetanus with thestandard application technique.The pain was evaluated with Number rating scale. The pain was evaluated immediately after vaccination and hemodynamic parameters were examined before and after the vaccination. A total of 32 pregnant women completed the study in the standard application group.
  Interventions: Procedure: Standard Injection technique

INTERVENTIONS:
Procedure: Helfer skin tap injection technique — 1. Place the patient in a seated position and open his right arm to inject into the deltoid muscle.
  2. After determining the injection site, use the tips of the dominant hand fingers to hit the skin (about 15 strokes) for about five seconds to soften the muscles.
  3. After cleaning the skin with alcohol, remove the syringe cover from the dominant hand. Make a V with the non-dominant hand and hit the skin three times.
  4. During the third stroke, prick the syringe into the muscle at 90 degrees angle at the same time.
  5. After aspiration, continue to hit the skin with the tips of the non-dominant hand fingers while injecting the drug with the dominant hand at a rate of 1 ml / 10 seconds.
  6. After injecting the drug, make the non-dominant hand V-shaped and hit the skin three times, pulling the syringe needle out at the same time during the third stroke
  Other Names: Helfer Skin Tap Group
  Arms: Helfer Skin Tap Group
Procedure: Standard Injection technique — 1. Place the patient in a seated position and open his right arm to inject into the deltoid muscle area.
  2. After determining the injection site, prepare the skin with alcohol.
  3. Grasp the skin with the thumb and index finger of the non-dominant hand and prick the syringe into the muscle at a 90-degree angle.
  4. After aspiration, inject the drug with the dominant hand at a rate of 1 ml /10 seconds.
  5. Remove the syringe needle 10 seconds after the drug is consumed
  Other Names: Standard Application Group
  Arms: Standard Application Group

SUMMARY:
Intramuscular (IM) vaccination administered using the right injection technique is known to cause less pain and injury. Nurses employ different approaches like applying pressure, tapping the skin, cold and hot applications for reducing the pain caused by the IM vaccine administration. Helfer skin tap is among the techniques that relax muscles.

The aim of the study was to determine the effect of Helfer skin tap technique on pain reduction and hemodynamic parameters during tetanus injection in pregnant women. This study was conducted on pregnant women who applied to the Family Health Center to get a tetanus vaccine. The Helfer skin tap and standard application groups each included 33 and 32 pregnant women, respectively.

DETAILED DESCRIPTION:
In 1988, Joanne Helfer developed the "Helfer Skin Tap Technique" which is applied by touching the skin over the injection site and attempted to reduce the intramuscular injection-related pain. In this technique, after determining the injection site, nearly 15 strokes are made on the skin for almost five seconds using the fingertips of the dominant hand in order to soften the muscles. Later, the skin is cleaned with alcohol, the non-dominant hand is put in V shape and the skin is hit three times. During the third stroke, the syringe is pricked into the muscle with a 90-degree angle at the same time. Making a few taps relaxes the muscles and counting to three helps synchronizing the muscle tap and injection and standardizes the technique. Mechanical stimulation of muscle fibers of larger diameters decreases the effect of smaller, pain generating fibers. According to the gate control theory suggested by Roger Metzack and Past Wall (1965), in addition to a mechanical stimulation during an IM injection, this technique also causes distraction, which, in turn, helps reducing pain.

The study aimed to determine the effect of Helfer skin tap technique on pain reduction and hemodynamic parameters during tetanus injection in pregnant women. This study was a randomized clinical trial conducted in Manisa Soma Family Health Center in Turkey. The study was conducted with 65 pregnant women who got tetanus vaccine. Tetanus vaccine was administered using the Helfer skin tap techniques to 33 of the pregnant women and standard IM injection technique to 32 women. The pain was evaluated immediately after vaccination and hemodynamic parameters were examined before and immediately after the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* being pregnant,
* having no infection, scar tissue, or incision, and receiving parenteral treatment in their injection area
* having no history of pain in their injection are
* applying for tetanus vaccine
* speaking Turkish
* voluntariness.

Exclusion Criteria:

* under the age of 18
* not being pregnant
* having a vaccination other than tetanus,
* having pain or a local infection prior to vaccination,
* having a circulatory disorder, peripheral vascular disease,
* cognitive and psychological problems,
* using painkillers at least 6 hours before the procedure,
* refusing to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Description of the pregnant women's demographics and clinical backgrounds. | It was implemented on the first day of the study and it took approximately 10-15 minutes to fill out the form.
  Questions about the pregnant women's descriptive characteristics such as age, education and employment status, Body Mass Index, smoking status, number of children and pregnancy, having intramuscular injection and any problem after intramuscular injection, and number of tetanus injection were asked using the questionnaire.
To evaluate peripheral oxygen saturation (%) immediately before tetanus vaccine in all women. | It was implemented immediately before tetanus vaccine administration in all women.
  Peripheral oxygen saturation (%) were evaluated immediately before tetanus vaccine administration in all women.
To evaluate heart rate (per minute) immediately before tetanus vaccine in all women. | It was implemented immediately before tetanus vaccine administration in all women.
  Heart rate (per minute) were evaluated immediately before tetanus vaccine administration in all women.
To evaluate respiratory rate (per minute) immediately before tetanus vaccine in all women. | It was implemented immediately before tetanus vaccine administration in all women.
  Respiratory rate (per minute) were evaluated immediately before tetanus vaccine administration in all women.
To evaluate systolic blood pressure (mm/Hg) and diastolic blood pressure (mm/Hg) immediately before tetanus vaccine in all women. | It was implemented immediately before tetanus vaccine administration in all women.
  Systolic blood pressure (mm/Hg) and diastolic blood pressure (mm/Hg) were evaluated immediately before tetanus vaccine administration in all women.

SECONDARY OUTCOMES:
To evaluate the pain level in the Helfer skin tap group with the Number rating scale in which 0 is defined as no pain and 10 as maximum pain. | It was implemented immediately after Tetanus vaccine that was administered using the Helfer skin tap techniques
  To evaluate the pain level immediately after Tetanus vaccine that was administered using the Helfer skin tap technique with the Number rating scale in which 0 is defined as no pain and 10 as maximum pain.
To evaluate the pain level in the Standart intramuscular injection group with the Number rating scale in which 0 is defined as no pain and 10 as maximum pain. | It was implemented immediately after Tetanus vaccine that was administered using the the Standart intramuscular injection techniques
  To evaluate the pain level immediately after Tetanus vaccine that was administered using the the Standart intramuscular injection with the Number rating scale in which 0 is defined as no pain and 10 as maximum pain.
To evaluate peripheral oxygen saturation (%) immediately after tetanus vaccine in all women. | It was implemented immediately after tetanus vaccine administration in all women
  Peripheral oxygen saturation (%) were evaluated immediately after tetanus vaccine administration in all women.
To evaluate heart rate (per minute) immediately after tetanus vaccine in all women. | It was implemented immediately after tetanus vaccine administration in all women
  Heart rate (per minute) were evaluated immediately after tetanus vaccine administration in all women.
To evaluate respiratory rate (per minute) immediately after tetanus vaccine in all women. | It was implemented immediately after tetanus vaccine administration in all women
  Respiratory rate (per minute) were evaluated immediately after tetanus vaccine administration in all women.
To evaluate systolic blood pressure (mm/Hg) and diastolic blood pressure (mm/Hg) immediately after tetanus vaccine in all women. | It was implemented immediately after tetanus vaccine administration in all women
  Systolic blood pressure (mm/Hg) and diastolic blood pressure (mm/Hg) were evaluated immediately after tetanus vaccine administration in all women.

CONTACTS AND LOCATIONS:
Overall Officials: Aslı Karakuş Selçuk, PhD, Principal Investigator — Manisa Celal Bayar University
Locations (1):
- Manisa Celal Bayar University, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No